CLINICAL TRIAL: NCT03680976
Title: Anti-Inflammatory Lipid Mediators in Asthma
Acronym: ALMA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study will not take place at the University of Pittsburgh
Sponsor: Sally E. Wenzel MD (Other)
Responsible Party: Sponsor-Investigator, Sally E. Wenzel MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRO16020149
Record Dates: First submitted 2016-03-09; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Asthma
Keywords: Asthma; Obesity; Nitrated fatty acids
MeSH Terms: conditions — Asthma; Obesity | interventions — CXA-10

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10-nitro-octadeca-9-enoic acid (CXA-10) (Experimental): CXA-10 150 mg tablet taken orally once a day for 12 weeks
  Interventions: Drug: CXA-10
- Placebo (Placebo Comparator): Placebo 150 mg tablet taken orally once a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CXA-10 — Liquid-filled capsule containing 150 mg CXA-10 in super refined olive oil.
  Other Names: 10-nitro-octadeca-9-enoic acid
  Arms: 10-nitro-octadeca-9-enoic acid (CXA-10)
Drug: Placebo — Liquid-filled capsule containing olive oil manufactured to mimic CXA-10 150 mg capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of 10-nitro-9(E)-octadec-9-enoic acid (CXA-10) in obese adult asthmatics. The study's hypothesis is that 150 mg/day of CXA-10 for 12 weeks will alleviate obesity-related airway hyper-reactivity in obese adult asthmatics.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate completion of informed consent process with written documentation. Male and female patients, 18 to 65 yrs old female subjects should be either post-menopausal, surgically sterile, or women of child-bearing potential (WOCP) with a negative pregnancy test prior to entering the study and who agree to use an acceptable method of contraception, for the duration of the study.
2. Diagnosis of asthma: based on previous physician diagnosis for > 6 months, and either baseline pre-bronchodilator (BD) FEV1 between 50 and 90% predicted with a 12% or greater bronchodilator response to 4 puffs of albuterol or PC20 methacholine (16 mg) if no BD response (<12% change), within 2 years of Visit 0. If no historical reversibility or historical PC20, and the participant does not reverse 12% at V0, the participant can return for V0a to meet this eligibility criteria.
3. Daily treatment with inhaled corticosteroids and long acting beta agonists (ICS/LABA) combination medication for at least 3 months; on a stable dose for the 4 weeks prior to Visit 0
4. Asthma control questionnaire ACQ > 1.5 & ≤ 3
5. Smoking history <10 pack years and no smoking in the last year
6. Body Mass Index (BMI) ≥ 30 kg/m2
7. Hemoglobin A1c (HbA1c) <8%
8. Average systolic blood pressure <160 or diastolic < 100 mmHg (average of three measurements))
9. Resting HR ≥45 beats per minute (BPM) after 5 minute rest at screening
10. QTcF interval (Fredericia's correction factor) must be ≤430 msec at screening and pre-dose for males and ≤450 msec for females.
11. For randomization: No exacerbations or treatment failures during the run in. Patients, who exacerbate or experience treatment failure during the run-in, may re-enroll 4 weeks after the exacerbation has resolved (completed course of systemic corticosteroids).

Exclusion Criteria:

1. Respiratory tract infection within the last 4 weeks
2. Oral or systemic corticosteroid burst within the last 4 weeks
3. Asthma-related hospitalization within the last 2 months
4. Three or more asthma exacerbations requiring treatment with systemic corticosteroids in the past year consistent with severe asthma
5. Asthma-related ER visit within the previous 4 weeks
6. Significant or uncontrolled concomitant medical illness including (but not limited to) heart disease, cancer, or diabetes at the discretion of the investigator
7. History of ICU admission/intubation due to asthma in the past year
8. Current statins use, patients may stop and re-enroll after 4 weeks of stopping statins
9. Positive pregnancy test at screening and at pre-dose
10. Women who are breastfeeding
11. Women of childbearing potential who are unwilling to use an acceptable method of birth control.
12. Intolerance or hypersensitivity to the CXA-10 or it's excipients
13. Treatment with any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to the beginning of dosing (this includes investigational formulations of marketed products, inhaled and topical drugs
14. Unable or unlikely to complete study assessments or the study intervention (i.e. bronchoscopy) poses undue risk to patient in the opinion of the Investigator;
15. Any kind of oral nitrates such as nitroglycerin
16. Any clinical history of cardiovascular events, arrhythmias, fainting, palpitations within the previous 3 years
17. Personal or family history of congenital prolonged QT syndromes or sudden unexpected death due to a cardiac reason
18. History of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions, with the exception of basal cell or squamous cell carcinomas of the skin
19. Cervical carcinoma in situ or other malignancies curatively treated and with no evidence of disease for at least 5 years
20. History of alcohol or drug abuse in the 6 month period prior to enrollment
21. Treatment with vitamins, herbal and dietary supplements within 7 days or 5 - ½ lives whichever is longer prior to dosing until the final study visit, whichever is longer prior to dosing until the final study visit. (may rescreen after a washout)
22. Resting heart rate ≥100 BPM after 5 minutes rest at screening
23. Subjects with any other clinically relevant ECG parameter abnormality (e.g., PR interval, QRS deviation) or any clinically significant ECG abnormality will be excluded from the study. Any clinically significant abnormalities on 12-lead ECG at screening including, but not limited to any of the following:

    * PR interval >200 msec or <120 msec
    * Non-specific intra-ventricular conduction delay (IVCD) with QRS duration ≥110 msec and where the morphology does NOT meet criteria for left (LBBB) or right bundle branch block (RBBB)
    * Incomplete RBBB as defined by QRS duration ≥110 msec but <120 msec with RBBB pattern
    * Complete RBBB and LBBB
    * Evidence of second- or third- degree AV block
    * Pathological Q-waves (Q-wave wider than 0.04 sec or depth greater than 0.4-0.5 mV)
    * Evidence of ventricular pre-excitation
    * Evidence of left axis deviation (left axis deviation is -30 to -90 degrees) but not normal leftward axis, ST-T wave abnormalities, LBBB and/or RBBB
24. Any clinically significant murmurs evident on auscultation of the heart (including evidence of mitral valve prolapse)
25. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3.0X upper limit of normal (ULN), gamma-glutamyl transferase (GGT) >3X ULN, and total bilirubin >2X ULN. If all liver function tests (LFTs) are within normal limits (WNL) and total bilirubin is elevated, examination of direct and indirect bilirubin may be conducted. Subjects with indirect total bilirubin up to 3X ULN are presumed to have Gilbert's syndrome and may be enrolled if all other LFTs are WNL
26. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures)
27. Diagnosis of HIV
28. Patients with multiple sclerosis on dimethyl fumarate (tecfidera)
29. Patients with asthma on biological therapy (i.e. mepolizumab, omalizumab)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in airway responsiveness after treatment with CXA-10 using a methacholine challenge test | 12 weeks
  Measured by the response to administration of methacholine. The PC20 is a calculated value of the amount of methacholine required to cause a 20% fall in the subject's FEV1.

SECONDARY OUTCOMES:
Treatment with CXA-10 compared to baseline: Change in the concentration of Nitrite/Nitrate (NO2/NO3). and NO2-Conjugated Linoleic Acid (CLA) in plasma and urine | 12 weeks
  Measured using analysis of plasma and urine at baseline and after treatment with CXA-10.
Treatment with CXA-10 compared to baseline: Characterization of the pharmacokinetic (PK) profile of CXA-10 in plasma and urine | 12 weeks
  Measured using analysis of plasma and urine at baseline and after treatment with CXA-10.
Treatment with CXA-10 compared to baseline: Changes in airway epithelial gene expression | 12 weeks
  Measured using bronchial samples from the subjects randomized to undergo a bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sally E Wenzel, MD, Principal Investigator — The University of Pittsburgh
Locations (1):
- The University of Pittsburgh Asthma Institute at UPMC, Pittsburgh, Pennsylvania, United States